CLINICAL TRIAL: NCT07034144
Title: Comparison of Chiropractic Diversified Technique and Drop Table Application in Patients With Neck Pain
Brief Title: Chiropractic Care for Neck Pain: Comparing Diversified Technique and Drop Table Method
Acronym: CDTDTM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SEFA HAKTAN HATIK (Other)
Responsible Party: Sponsor-Investigator, SEFA HAKTAN HATIK, Asst. Professor, Sinop University
Organization: Sinop University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMT0007
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Spinal Manipulation; Neck Pain; Non Specific Neck Pain; Chiropractic
Keywords: Chiropractic; Neck pain; Drop Table; Spinal Manipulation
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This study is designed as a double-blind, randomized controlled trial involving three groups: the Diversified technique group, the Drop Table application group, and a control group. Although the nature of manual therapy prevents complete blinding of participants, all were only informed that they would receive chiropractic care, without specifying the technique applied. Thus, participants were blinded to the specific intervention type. The practitioners administering the treatments were not blinded due to the need to apply the appropriate technique. However, all outcome assessments were performed by an independent evaluator who was blinded to group allocation and not involved in the intervention process, ensuring objective measurement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diversified Group (Experimental): Participants in this group will receive chiropractic treatment using the Diversified Technique.
  The intervention will be applied twice per week for 4 weeks by a chiropractor. The treatment will focus on cervical spine adjustments targeting areas of joint dysfunction associated with mechanical neck pain.
  Each session will last approximately 20 minutes. Standardized protocols will be followed to ensure consistency.
  Interventions: Other: Cervical Spine Manipulation
- Drop Table Group (Experimental): Participants in this group will receive chiropractic treatment using the Drop Table Technique.
  The intervention will be applied twice per week for 4 weeks by a chiropractor. The treatment will involve high-velocity, low-amplitude thrusts delivered with the assistance of a segmented drop table designed to reduce resistance and enhance precision during spinal adjustments.
  The focus will be on the cervical spine region related to mechanical neck pain. Each session will last approximately 20 minutes, following standardized protocols to ensure treatment consistency.
  Interventions: Other: Drop Table Technique
- Control Group (No Intervention): This group did not undergo any interventions.

INTERVENTIONS:
Other: Drop Table Technique — The Drop Table Technique is a chiropractic intervention that utilizes a segmented treatment table with adjustable sections that can be elevated slightly and then dropped.
  During the procedure, a high-velocity, low-amplitude (HVLA) thrust is applied while the specific segment of the table drops slightly in coordination with the thrust.
  This technique aims to reduce the resistance experienced during the adjustment and to enhance the mechanical effect on targeted spinal joints.
  In this study, the Drop Table Technique will be specifically applied to the cervical spine to address mechanical neck pain.
  All applications will be performed by a licensed chiropractor using standardized positioning and adjustment protocols to ensure consistency across sessions.
  Arms: Drop Table Group
Other: Cervical Spine Manipulation — Cervical spinal manipulation (SM) will be applied with the participant supine to restrictions found on motion palpation, following the technique described by Bergmann and Peterson. The participant's head and neck will be simultaneously rotated and laterally flexed over the contact point-specifically, the posterior supramastoid groove or zygomatic arch (C0-C1), the posterior aspect of the transverse process (C1-C2), or the posterior articular pillar of superior vertebrae (C2-C7)-to the end of passive range of motion (ROM).
  Subsequently, a high-velocity, low-amplitude thrust will be delivered in the direction of restricted movement. Participants with greater ROM restriction in the lateral plane will receive more laterally-to-medially directed thrusts. Participants with more restriction in rotation will be given thrusts in the direction of restricted axial rotation, and those with more restriction in extension will receive more anteriorly directed thrusts.
  Arms: Diversified Group

SUMMARY:
This study aims to compare the effects of two different chiropractic techniques, Diversified and Drop Table, on pain levels, cervical joint range of motion, and neck muscle strength in individuals with non-specific neck pain.

DETAILED DESCRIPTION:
This randomized controlled trial aims to compare the effectiveness of two chiropractic techniques - the Diversified Technique and the Drop Table Technique - in individuals with mechanical neck pain. Mechanical neck pain is a common musculoskeletal condition associated with impaired cervical mobility, pain, and reduced quality of life.

Participants will be randomly assigned to one of three arms: (1) Diversified Technique group, (2) Drop Table Technique group, and (3) control group with no intervention. The interventions will be administered twice per week for four weeks by a chiropractor following standardized protocols. All participants will undergo evaluations at baseline and at the end of the 4-week intervention period.

The primary outcome measure is pain intensity and quality, assessed using the full version of the McGill Pain Questionnaire (MPQ), which evaluates sensory, affective, and evaluative components of pain. Secondary outcomes include cervical range of motion (CROM) and isometric neck muscle strength, measured with a goniometer and handheld dynamometer, respectively.

This study seeks to provide evidence on the comparative clinical effectiveness of two widely used chiropractic techniques for neck pain management. The findings may guide clinicians in selecting appropriate manual therapy approaches for patients with non-specific mechanical neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Sign a voluntary informed consent form.
* Be between 18 and 65 years of age.
* Have previously consulted an orthopedist or physical therapist for neck pain.
* Have no contraindications to chiropractic interventions.
* Have no history of cervical surgery.
* Report neck pain lasting longer than 7 days.

Exclusion Criteria:

* Are under 18 or over 65 years of age.
* Have experienced cervical trauma within the last month.
* Have any systemic illness.
* Have any contraindication for chiropractic intervention (e.g., brain tumor, cervical fracture).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06-14 (Estimated); Primary Completion 2025-07-14 (Estimated); Study Completion 2025-08-14 (Estimated)

PRIMARY OUTCOMES:
McGill Pain Questionnaire (MPQ) | Baseline and Week 4
  Pain will be assessed using the full version of the McGill Pain Questionnaire (MPQ), which evaluates both the sensory, affective, evaluative, and miscellaneous components of pain.
  The MPQ includes:
  A list of 78 pain descriptors grouped into 20 categories, The Pain Rating Index (PRI), derived from the sum of rank values for selected descriptors, A Present Pain Intensity (PPI) score, rated on a scale of 0 (no pain) to 5 (excruciating), A Visual Analog Scale (VAS) for overall pain intensity. The primary outcome will be the change in total PRI and PPI scores from baseline to the end of the 4-week intervention.
  Measure Type:
  Ordinal and Continuous (PRI: rank-based score; PPI: 0-5 scale)
  Unit of Measure:
  Score (no unit)

SECONDARY OUTCOMES:
Cervical Range of Motion | Baseline and 4th week
  Measured in degrees using a goniometer in all planes of cervical motion.
Isometric Neck Muscle Strength | Baseline and 4th week
  Isometric neck muscle strength in flexion, extension, and right and left lateral flexion will be manually assessed using a microFET2 handheld dynamometer (Hoggan Health Industries).

CONTACTS AND LOCATIONS:
Overall Officials: SEFA H HATIK, Asst. Prof., Principal Investigator — Sinop University
Locations (1):
- Sinop University, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No